CLINICAL TRIAL: NCT07361263
Title: Plasma Oxytocin in Response to Oral Estradiol Valerate and Ethinylestradiol in Healthy Controls and Patients With AVP-Deficiency
Brief Title: Plasma Oxytocin Response to Oral Estrogens in Healthy Controls and AVP-Deficiency
Acronym: PHOENIX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2025-02197;kt25ChristCrain5
Record Dates: First submitted 2026-01-05; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: AVP Deficiency; Diabetes Insipidus
Keywords: Oxytocin; estradiol valerate; ethinylestradiol
MeSH Terms: conditions — Diabetes Insipidus, Neurogenic; Diabetes Insipidus | interventions — Estradiol

STUDY DESIGN:
Intervention Model Description: This study will be conducted in two parts. Part 1 is a double-blinded, randomized cross-over proof-of-concept trial in healthy adults. Part 2 is an open-labeled single arm pilot study in adults with an established diagnosis of AVP-Deficiency. Study parts 1 and 2 will be conducted consecutively.
  For part 1 16 participants will be enrolled and for part 2 12 patients will be enrolled.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- estradiol valerate (Experimental)
  Interventions: Drug: estradiol valerate
- esthinylestradiol (Experimental)
  Interventions: Drug: esthinylestradiol

INTERVENTIONS:
Drug: estradiol valerate — estradiol valerate
  Arms: estradiol valerate
Drug: esthinylestradiol — estradiol valerate
  Arms: esthinylestradiol

SUMMARY:
The PHOENIX study aims to investigate whether oral estradiol valerate (EV) and ethinylestradiol (EE) can stimulate oxytocin (OXT) and neurophysin-1 (NP-1) release in humans. The goal is to assess their potential as a safe diagnostic stimulation test for oxytocin deficiency, particularly in patients with arginine vasopressin (AVP) deficiency.

DETAILED DESCRIPTION:
Oxytocin (OXT) and arginine vasopressin (AVP) are hypothalamic peptides involved in water balance and emotional regulation. Patients with AVP-Deficiency (central diabetes insipidus) often experience psychological symptoms such as anxiety and depressed mood, possibly due to coexisting OXT deficiency. Previous research showed that 3,4-Methylenedioxy-N-methylamphetamine (MDMA) can increase plasma OXT in healthy individuals but not in AVP-deficient patients, suggesting a clinically relevant OXT deficiency. However, the side effects of MDMA limit its clinical use as a diagnostic tool. Estrogen is known to stimulate OXT release via estrogen receptor β in the hypothalamus. This study evaluates whether oral estradiol valerate (EV) and ethinylestradiol (EE) can safely and effectively provoke OXT and NP-1 release, offering a potential alternative to MDMA-based tests.

The study consists of two parts:

Part 1 (Proof of Concept): A randomized, double-blind, cross-over trial in healthy adults to compare the stimulatory effects of EV and EE on plasma OXT and NP-1.

Part 2 (Pilot Study): An open-label trial in patients with AVP-Deficiency using the estrogen compound identified as most effective in Part 1, to determine whether OXT and NP-1 responses are blunted compared to healthy controls.

ELIGIBILITY:
Inclusion Criteria:

Part 1

1. Adult healthy controls
2. No medication (including hormonal contraception)
3. Female patients (except post-menopausal): regular cycle (21-35 days of duration) in the last 6 months

Part 2

1. Confirmed diagnosis of AVP-Deficiency
2. Age ≥ 18 years
3. Female patients (except post-menopausal): regular cycle (21-35 days of duration) in the last 6 months or in the case of hormone replacement therapy, with a 1-week pause from the respective treatment

Exclusion Criteria:

Part 1

1. Participation in a trial with investigational drugs within 30 days
2. BMI >30
3. Age >50
4. Illicit substance use (except for cannabis) during the last 30 days
5. Consumption of alcoholic beverages >15 drinks/week
6. Tobacco smoking >10 cigarettes/day
7. Pregnancy and breastfeeding
8. Hormonal contraception
9. Migraine with and without aura
10. Any cardiometabolic, cardiovascular, and hematological diseases (including deep vein thrombosis/pulmonary embolism and thrombophilia (DVT/PE))
11. Active liver dysfunction or alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) levels 2.5 times above the normal range
12. Diagnosed chronic kidney disease (CKD) > grade III (GRF < 30ml/min)

Part 2

1. Participation in a trial with investigational drugs within 30 days
2. BMI >30
3. Age >50
4. Illicit substance use (except for cannabis) during the last 30 days
5. Consumption of alcoholic beverages >15 drinks/week
6. Tobacco smoking >10 cigarettes/day
7. Pregnancy and breastfeeding
8. Hormonal contraception
9. Migraine with and without aura
10. Any cardiometabolic, cardiovascular, and hematological diseases (including DVT/PE and Thrombophilia)
11. Active liver dysfunction or alanine aminotransferase (ALAT) or aspartate aminotransferase (ASAT) levels 2.5 times above the normal range
12. Diagnosed CKD > grade III (GRF < 30ml/min)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-01-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Relative Change in Plasma Oxytocin | From baseline (0 min) to 300 minutes post-dose.
  The primary endpoint is the relative change in plasma oxytocin (OXT) concentrations (pg/mL respectively pM) from baseline to the maximum observed value within 300 minutes after administration of oral estradiol valerate (EV) or ethinylestradiol (EE). Baseline is defined as 100% of the initial pre-dose concentration.
Relative Change in Neurophysin-1 | From baseline (0 min) to 300 minutes post-dose.
  The primary endpoint is the relative change in neurophysin-1 (NP-1) concentrations (pg/mL respectively pM) from baseline to the maximum observed value within 300 minutes after administration of oral estradiol valerate (EV) or ethinylestradiol (EE). Baseline is defined as 100% of the initial pre-dose concentration.

SECONDARY OUTCOMES:
Area Under the Curve (AUC) for Plasma OXT and NP-1 | From baseline (0 min) to 300 minutes post-dose.
Peak change in plasma OXT/NP-1 levels | From baseline (0 min) to 300 minutes post-dose.
Time course of plasma OXT/NP-1 levels | From baseline (0 min) to 300 minutes post-dose.
Changes in Coagulation Parameters: time course (von Willebrand factor) | From baseline (0 min) to 300 minutes post-dose.
  Time course and peak of coagulation marker von Willebrand factor
Changes in Coagulation Parameters: time course (Protein S) | From baseline (0 min) to 300 minutes post-dose.
  Time course and peak of coagulation marker Protein S
Changes in Coagulation Parameters: time course (D-dimer) | From baseline (0 min) to 300 minutes post-dose.
  Time course and peak of coagulation marker D-dimer
Changes in Coagulation Parameters: time course (Factor VIII) | From baseline (0 min) to 300 minutes post-dose.
  Time course and peak of coagulation marker Factor VIII
Changes in Coagulation Parameters: time course (Fibrinogen) | From baseline (0 min) to 300 minutes post-dose.
  Time course and peak of coagulation marker Fibrinogen
Changes in Coagulation Parameters: peak (von Willebrand factor) | From baseline (0 min) to 300 minutes post-dose.
  Peak of coagulation marker von Willebrand factor
Changes in Coagulation Parameters: peak (Protein S) | From baseline (0 min) to 300 minutes post-dose.
  Peak of coagulation marker Protein S
Changes in Coagulation Parameters: peak (D-dimer) | From baseline (0 min) to 300 minutes post-dose.
  Peak of coagulation marker D-dimer
Changes in Coagulation Parameters: peak (Factor VIII) | From baseline (0 min) to 300 minutes post-dose.
  Peak of coagulation marker Factor VIII
Changes in Coagulation Parameters: peak (Fibrinogen) | From baseline (0 min) to 300 minutes post-dose.
  Peak of coagulation marker Fibrinogen
Changes in Other Endocrine Hormones | From baseline (0 min) to 300 minutes post-dose.
  Time course of plasma estrogen, testosterone, copeptin, cortisol,Luteinizing Hormone/Follicle-Stimulating Hormone (LH/FSH), and other pituitary hormones.
Subjective Emotional Effects | At baseline (0 min), 30, 60, 90, 120, 150, 180, 210, 240, 270 and 300 minutes and 24 hours post-dose.
  Changes in subjective feelings assessed by Numeric Rating Scale (NRS). NRS will be repeatedly used to assess subjective alterations in consciousness over time. NRS will be presented as a range from 0 to 10 marked with "not at all" on the left and "extremely" on the right. The following NRS will be used: "any effect", "good effect", "bad effect", "liking", "high", "happy", "fear", "stimulated", "feeling close to others", "concentration", "thinking", "open", and "trust".
Adverse effects | 300 minutes post-dose.
  Participants will be asked to report any adverse events that occur during the sessions or between sessions at the start of the next session. The test requires about 2 minutes.
List of complaints (LC) | 300 minutes post-dose.
  The LC consists of 66 items, yielding a global score measuring physical and general discomfort. The LC list is administered at the beginning and the end of the session with reference to complaints throughout the entire session.
Changes in anxiety assessed by State-Trait Anxiety Inventory (STAI-State and Trait). | Baseline, 90 and 270 minutes post-dose.
  This is a questionnaire given to adults to determine the general anxiety levels. Based on responses to 20 items, with scores ranging from 1 ("almost never") to 4 ("almost always"), a total score is calculated. The total trait score (STAI-T) ranges from 20 to 80, with higher scores indicating more pronounced anxiety and scores. The STAI-T evaluates relatively stable aspects of "anxiety proneness," including general states of calmness, confidence, and security. A score above 45/80 indicating clinically significant anxiety symptoms. The state score (STAI-S) evaluates the current state of anxiety, asking how respondents feel "right now," using items that measure subjective feelings of apprehension, tension, nervousness, worry, and activation/arousal of the autonomic nervous system. We will use the STAI-T for the baseline visit and the STAI-S for the treatment visits. The test requires about 5 minutes.
Emotion Recognition Performance - EmBody/EmFace Task | Baseline and 270 minutes post-dose.
  The EmBody and EmFace subtasks comprise each of 42 stimuli showing body or facial expressions of angry, happy, or neutral affect (14 clips per emotion, half in front view and half in half-profile side view from the left). Stimuli last 1.5 seconds at 24 frames per second and are geometrically and optically standardized to prevent biases induced by ethnic cues (e.g., hair or skin tone) or clothing. Item order is pseudorandom to prevent sequence effects and was determined using the following constraints: the same emotion is shown no more than twice in a row; the same view per emotion is not shown consecutively (i.e., no angry-front, angry-front). The test is performed twice during each treatment visit.
Emotion Recognition Performance - Face Recognition Task (FERT) | At 270 minutes post-dose.
  The FERT is used to assess recognition of basic emotions. The task includes 10 neutral faces and 160 faces that express one of four basic emotions (i.e., happiness, sadness, anger, and fear), with pictures morphed between 0% (neutral) and 100% in 10% steps. Two female and two male pictures are used for each of the four emotions. Stimuli are shown in random order for 500 ms and are then replaced by the rating screen where participants have to indicate the correct emotion. The outcome measure is accuracy (proportion correct). The test data is recorded on a computer and processed into scores for each emotion using an established matlab routine according to standard operating procedures (SOP) (clinical pharmacology, Orca DKF). The test is performed once during each treatment visit, exactly 270min after EV/EE administration.
Vital parameters: blood pressure | 30 minutes pre-dose; 0, 30, 60, 120, 150, 180, 210, 240, 270, 300minutes, 24hours post-dose.
  Blood pressure (systolic and diastolic) will be measured at several timepoints during the treatment visit
Vital parameters: heart rate | 30 minutes pre-dose; 0, 30, 60, 120, 150, 180, 210, 240, 270, 300minutes, 24hours post-dose.
  Heart rate will be measured at several timepoints during the treatment visit
Vital parameters: body temperature | 30 minutes pre-dose; 0, 30, 60, 120, 150, 180, 210, 240, 270, 300minutes, 24hours post-dose.
  body temperature will be measured at several timepoints during the treatment visit
Concentration of Plasma Sodium | At 0, 180 and 300 minutes post-dose.
  Sodium concentration (mmol/l) will be assessed in plasma.
Concentration of Plasma Potassium | At 0, 180 and 300 minutes post-dose.
  Sodium concentration (mmol/l) will be assessed in plasma.
Concentration of Saliva Oxytocin | At 0, 60, 90, 120, 180, 270, 300 minutes and 24 hours post-dose.

CONTACTS AND LOCATIONS:
Overall Officials: Mirjam Christ-Crain, Prof. Dr., Study Chair — University Hospital of Basel
Locations (1):
- University Hospital Basel, Basel, Switzerland